CLINICAL TRIAL: NCT03407807
Title: Isolated Fetal Splenic Cyst : Prenatal Diagnosis and Postnatal Evolution
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0331
Record Dates: First submitted 2017-10-25; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-10

CONDITIONS: Pregnant Women
Keywords: Fetal Splenic cyst; Differential Diagnosis; Evolution and complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to describe prevalence, radiologic and ultrasound evolution during pregnancy, postnatal evolution and treatment strategy in case of isolated fetal spelnic cyst

DETAILED DESCRIPTION:
The aim of this study was to describe prevalence, radiologic and ultrasound evolution during pregnancy, postnatal evolution and treatment strategy in case of isolated fetal spelnic cyst. The investigators performed a retrospective study in the Montpellier Prenatal Diagnosis Centre between 2007 and 2017. All pregnant women referred to this unit after routine ultrasound examination with a suspected splenic cyst were included. Participant all benefit a reference ultrasound to perform a detailed morphological examination. In any doubt about diagnosis, a MRI exam wad proposed. Then patient were followed regularly. At birth, all newborn babys had medical examination to search early complication. Then, children had a surgical consultation and regular ultrasound examinations were performed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnent women with an isolated suspected fetal splenic cyst between 2007 and 2017 in Montpellier Prenatal Diagnosis Center

Exclusion Criteria:

* All others fetal diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnent women with an isolated suspected fetal splenic cyst
Sampling Method: Probability Sample
Enrollment: 5450 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Prenatal ultrasound evolution of fetal splenic cysts during pregnancy | 1 day
  Prenatal ultrasound evolution of fetal splenic cysts during pregnancy: persistence, increasing/decreasing in size, disappearance

SECONDARY OUTCOMES:
Prenatal Magnetic Resonance imaging (MRI) evolution of fetal splenic cyst | 1 year
  Prenatal Magnetic Resonance imaging (MRI) evolution of fetal splenic cyst (persistence, increasing/decreasing in size, disappearance)
Post natal ultrasound evolution at birth of the cyst | 1 year
  Post natal ultrasound evolution at birth of the cyst : persistence, increasing/decreasing in size, disappearance
Post natal MRI evolution at birth of the cyst | 1 year
  Post natal MRI evolution at birth of the cyst : persistence, increasing/decreasing in size, disappearance
1 year ultrasound evolution of the cyst | 1 year
  1 year ultrasound evolution of the cyst : persistence, increasing/decreasing in size, disappearance
1 year MRI evolution of the cyst | 1 year
  1 year MRI evolution of the cyst : persistence, increasing/decreasing in size, disappearance

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France